CLINICAL TRIAL: NCT04642040
Title: Effectiveness of Pulmonary Rehabilitation Program in Patients With SARS-CoV-2 Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Enes Efe Is, MD, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2857
Record Dates: First submitted 2020-11-21; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Covid19 Pneumonia; SARS-CoV 2 Pneumonia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Rehabilitation (Experimental): Patients are included in a personalized pulmonary telerehabilitation program consisting of patient education, respiratory and peripheral muscle training, and breathing strategies for 4 weeks. In the telerehabilitation program, exercises will be supervised by a physiotherapist two days a week, and patients will be asked to do the exercises themselves for the other 3 days. Patients will also receive instructional exercise videos for these 3 days.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Positioning,breathing techniques (diaphragmatic breathing, alternate breathing, and pursed-lip breathing),respiratory muscle exercises, joint ROM exercises, early-mobilization and progressive ambulation, peripheral muscle strengthening exercises

SUMMARY:
The aim of the study is to investigate the efficacy of pulmonary rehabilitation (PR) program to patients with Sars-CoV-2 pneumonia in the post-acute period on pulmonary functions, exercise capacity and anxiety level.

100 patients diagnosed with Sars-CoV-2 pneumonia will be enrolled in this prospective, interventional study according to inclusion/exclusion criteria. Patients will be evaluated and a personalized PR program will be organized before hospital discharge. After discharge, the pulmonary rehabilitation program will continue in telerehabilitation.

In the telerehabilitation program, exercises will be supervised by a physiotherapist two days a week, and patients will be asked to do the exercises themselves for the other 3 days. Patients will also receive exercise videos for these 3 days.

Patients will be followed for 4 weeks and will be called for final evaluation

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia without having severe findings or a need for oxygen support therapy (mild pneumonia) accompanying special conditions (chronic lung / heart disease / diabetes / hypertension / neuromuscular disease history / elderly / immobility etc.)
* Severe pneumonia (A suspicion of fever or respiratory tract infection and having one accompanying finding: respiration rate >30/min; severe respiratory distress; or SpO2 ≤93% in ambient air.) cases after they get clinically stable (decreased fever, reduced dyspnea, respiratory rate 90%)
* At least 7 days since the diagnosis of SARS-CoV-2 in order to reduce the viral load and the risk of transmission
* Being able to make video calls for telerehabilitation

Exclusion Criteria:

* Serious cardiovascular, cerebrovascular, neuromuscular and other systemic diseases that affect physical activity
* Psychiatric illness and cognitive deficit that will affect patient's exercise cooperation
* Pregnancy
* The deterioration in the general condition of the patient, worsening of the lung findings
* Acute respiratory distress syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in Dyspnea level as measured by modified Medical Research Council (mMRC) Dyspnea Scale | 4 weeks
  The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4. 0: no breathlessness except on strenuous exercise; 4: too breathless to leave the house, or breathless when dressing or undressing.
Change in functional capacity as measured by 30-second sit-to-stand test | 4 weeks
  30 sec- STS determines lower extremity strength and physical fitness in older adults. The number of repetitions is recorded.

SECONDARY OUTCOMES:
Change in physical activity level as measured by International Physical Activity Questionnaire (IPAQ) -Short Form | 4 weeks
  IPAQ-Short Form is used to measure level of physical activity.It consists of 7 questions that provide information about time spent on walking, moderate to vigorous physical activities, and time spent sitting. The energy required for the activities was calculated by the MET-minute/week score. Standard MET values for these activities are: Walking = 3,3 METS; Moderate Physical Activity = 4,0 METS; Vigorous Physical Activity = 8.0 METS; Sitting = 1,5 METS
Change in anxiety and depression as measured by Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression.The total scores range is 0-21 for both depression and anxiety scores. A higher score indicates a worse depression and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sahillioglu, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital PMR Clinic
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtais Aytur Y, Koseoglu BF, Ozyemisci Taskiran O, Ordu-Gokkaya NK, Unsal Delialioglu S, Sonel Tur B, Sarikaya S, Sirzai H, Tekdemir Tiftik T, Alemdaroglu E, Ayhan FF, Duyur Cakit BD, Genc A, Gundogdu I, Guzel R, Demirbag Karayel D, Bilir Kaya B, Oken O, Ozdemir H, Soyupek F, Tikiz C. Pulmonary rehabilitation principles in SARS-COV-2 infection (COVID-19): A guideline for the acute and subacute rehabilitation. Turk J Phys Med Rehabil. 2020 May 12;66(2):104-120. doi: 10.5606/tftrd.2020.6444. eCollection 2020 Jun. PMID 32760887